CLINICAL TRIAL: NCT01199588
Title: A Randomized, Parallel Group, Dose-Ranging, Controlled, Multi-Center Study to Assess the Efficacy and Safety of Nexagon® in the Treatment of Subjects With a Venous Leg Ulcer
Brief Title: A Study to Investigate the Efficacy, Safety and Tolerability of Nexagon® as a Topical Treatment for Subjects With Venous Leg Ulcers
Acronym: NOVEL2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OcuNexus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEX-ULC-007
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Venous Leg Ulcers
Keywords: VLU; Venous Leg Ulcers; Ulcers; chronic wounds; wounds; Nexagon; CoDa
MeSH Terms: conditions — Ulcer; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nexagon® High Dose (Experimental): Weekly applications of Nexagon® high dose in addition to compression dressings.
  Interventions: Drug: Nexagon® High Dose
- Nexagon® Vehicle (Placebo Comparator): Weekly applications of Nexagon® Vehicle in addition to compression dressings.
  Interventions: Drug: Nexagon® Vehicle
- No Investigational Product (No Intervention): Weekly application of compression dressings.
- Nexagon® Low Dose (Experimental): Weekly applications of Nexagon® low dose in addition to compression dressings.
  Interventions: Drug: Nexagon® Low Dose

INTERVENTIONS:
Drug: Nexagon® Low Dose — Weekly, topical application of Nexagon® low dose used with compression dressings.
  Arms: Nexagon® Low Dose
Drug: Nexagon® High Dose — Weekly, topical application of Nexagon® high dose used with compression dressings.
  Arms: Nexagon® High Dose
Drug: Nexagon® Vehicle — Weekly, topical application of Nexagon® Vehicle used with compression dressings.
  Arms: Nexagon® Vehicle

SUMMARY:
This study is for subjects with a venous leg ulcer. The study is being done to determine if NEXAGON plus compression bandaging is more effective that placebo plus compression bandaging.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of venous leg ulceration supported by venous duplex ultrasonography demonstrating venous reflux > 0.5 seconds
2. Ankle brachial index of > 0.80
3. Venous Leg Ulcer (VLU) area greater than 2 cm2 and less than 20 cm2
4. Compliant with and able to tolerate high compression bandaging
5. VLU present for > 30 days prior to study entry
6. VLU is full thickness
7. The subject is willing and able to give informed consent

Exclusion Criteria:

1. Decrease or increase in the ulcer surface area by more than 40% during the 14 day run-in period
2. More than 75% of the VLU is on or below the malleolus
3. Presence of a non-study ulcer within 1.5 cm of the VLU
4. A VLU which shows signs of clinical infection or has cellulitis
5. The VLU wound bed has exposed bone, tendon or fascia
6. BMI > 45.0 kg/m2
7. Subject is not ambulatory
8. Subjects who have a past or present disease that, which as judged by the Investigator, may affect the safety of the subject or the outcome of the study
9. Cancerous cells in the VLU
10. HbA1c >10%
11. Blood biochemistry >3x upper limit of normal
12. Heart failure NYHA class III or IV
13. Subjects on renal replacement therapy
14. Immunocompromized subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Surface area reduction | 10 weeks

SECONDARY OUTCOMES:
Incidence of complete closure | 10 weeks
Time to complete closure | 10 weeks
Incidence of ulcer recurrence | 12 weeks post closure
Pain | 10 weeks
Incidence of adverse events | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tom Serena, MD, Principal Investigator — Penn North Centers For Advanced Wound Care, PA, USA
Locations (34):
- United States (21):
  - Associated Foot and Ankle Specialists, LLC, Phoenix, Arizona
  - Aung Foot Health Clinics, Tucson, Arizona
  - Southern Arizona Limb Salvage Alliance, Tucson, Arizona
  - Bay Area Foot Care, Castro Valley, California
  - Diabetic Foot & Wound Treatment Center, El Centro, California
  - Advanced Foot Care and Clinical Research Center, Fresno, California
  - Doctor's Research Network, South Miami, Florida
  - South Florida Wound Care Group, Tamarac, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Passavant Area Hospital, Jacksonville, Illinois
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Oceana Country Foot and Ankle, Toms River, New Jersey
  - St Luke's - Roosevelt Hospital Center Department of Surgery, New York, New York
  - Stonybrook Univeristy Medical Center, New York, New York
  - St. John Wound Center, Tulsa, Oklahoma
  - Penn North Center For Advanced Wound Care, Erie, Pennsylvania
  - Penn North Center For Advanced Wound Care, Kittaning, Pennsylvania
  - Center For Advanced Wound Care, Wyomissing, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Saint Paul's Women's Center, Dallas, Texas
  - DRMC Wound Clinic, Saint Geroge, Utah
- Australia (2):
  - South Sydney Vascular Centre, Sydney, New South Wales
  - Heidelberg Repatriation Hospital, Melbourne, Victoria
- New Zealand (2):
  - Awhinatina Health, Manukau, Auckland
  - Dunedin Hospital, Dunedin, Otago
- South Africa (9):
  - Dr D. Lakha, Johannesburg, Gauteng
  - Josha Research, Bloemfontein
  - Boland Ethical Research Group, Cape Town
  - Randles Road Medical Centre, Durban
  - Unitas Hospital, Johannesburg
  - WorthwhileClinical Trials, Johannesburg
  - Sunninghill Hospital, Johannesburg
  - Witwatersrand University Medical School, Johannesburg
  - GCT Mercantile Clinical Trial Centre, Port Elizabeth